CLINICAL TRIAL: NCT03194867
Title: A Phase 1/2 Study to Evaluate Safety, Pharmacokinetics and Efficacy of Isatuximab in Combination With Cemiplimab in Patients With Relapsed/Refractory Multiple Myeloma
Brief Title: Isatuximab in Combination With Cemiplimab in Relapsed/Refractory Multiple Myeloma (RRMM) Patients
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TCD14906; 2017-001431-39 (EudraCT Number); U1111-1189-4706 (Other: UTN)
Record Dates: First submitted 2017-06-19; First posted 2017-06-21 (Actual); Results first posted 2024-06-14 (Actual); Last update posted 2024-06-14 (Actual); Status verified 2024-05

CONDITIONS: Plasma Cell Myeloma
Keywords: Anti-CD38 monoclonal antibody
MeSH Terms: conditions — Multiple Myeloma | interventions — isatuximab; cemiplimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Isatuximab/cemiplimab (Regimen 1) (Experimental): Isatuximab on Days 1, 8, 15, and 22, then Days 1 and 15 in 28-day cycles up to disease progression.
  Cemiplimab on Days 1 and 15 in 28-day cycle up to disease progression.
  Interventions: Drug: Isatuximab SAR650984; Drug: Cemiplimab REGN2810
- Isatuximab/cemiplimab (Regimen 2) (Experimental): Isatuximab on Days 1, 8, 15, and 22, then Days 1 and 15 in 28-day cycles up to disease progression.
  Cemiplimab on Day 1 in 28-day cycle up to disease progression.
  Interventions: Drug: Isatuximab SAR650984; Drug: Cemiplimab REGN2810
- Isatuximab (Active Comparator): Isatuximab on Days 1, 8, 15 and 22, then Day 1 and 15 in 28-day cycles up to disease progression.
  Interventions: Drug: Isatuximab SAR650984

INTERVENTIONS:
Drug: Isatuximab SAR650984 — Pharmaceutical form: solution for infusion
  Route of administration: intravenous
  Other Names: Sarclisa
Drug: Cemiplimab REGN2810 — Pharmaceutical form: solution for infusion
  Route of administration: intravenous
  Arms: Isatuximab/cemiplimab (Regimen 1); Isatuximab/cemiplimab (Regimen 2)

SUMMARY:
Primary Objectives:

* To evaluate the safety and tolerability of the combination of isatuximab (also known as SAR650984) and cemiplimab (also known as REGN2810) in patients with relapse/refractory multiple myeloma.
* To compare the overall response of the combination of isatuximab and cemiplimab versus isatuximab alone in patients with RRMM based on International Myeloma Working Group (IMWG) criteria.

Secondary Objectives:

* To evaluate the efficacy as assessed by clinical benefit rate (CBR), duration of response (DOR), time to response (TTR), progression free survival (PFS), and overall survival (OS).
* To assess the pharmacokinetics (PK) of isatuximab and cemiplimab when given in combination.
* To assess the immunogenicity of isatuximab and cemiplimab when given in combination.

DETAILED DESCRIPTION:
The duration of the study for a patient will include a period for screening of up to 21 days and 3-month post treatment follow up. The cycle duration is 28 days. Patients will continue treatment until disease progression, unacceptable adverse events, consent withdrawal, or any other reason.

ELIGIBILITY:
Inclusion criteria:

* Patients must have a known diagnosis of multiple myeloma with evidence of measurable disease, as defined below:

  * Serum M-protein ≥1 g/dL (≥0.5 g/dL in case of immunoglobulin A [IgA] disease), AND/OR
  * Urine M-protein ≥200 mg/24 hours, OR
  * In the absence of measurable M-protein, serum immunoglobulin free light chain ≥10 mg/dL, and abnormal serum immunoglobulin kappa lambda free light chain ratio (<0.26 or >1.65).
* Patients must have received prior treatment with an immunomodulatory drug (IMiD) (for ≥2 cycles or ≥2 months of treatment) and a proteasome inhibitor (PI) (for ≥2 cycles or ≥2 months of treatment).
* Patients must have received at least 3 prior lines of therapy (Note: Induction therapy and stem cell transplant ± maintenance will be considered as one line).
* Patient must have achieved MR or better with any anti-myeloma therapy (ie, primary refractory disease is not eligible).

Exclusion criteria:

* Prior exposure to isatuximab or participated clinical studies with isatuximab.
* Prior exposure to any agent (approved or investigational) that blocks the programmed cell death-1 (PD-1)/PD-L1 pathway.
* Evidence of other immune related disease/conditions.
* History of non-infectious pneumonitis requiring steroids or current pneumonitis; history of the thoracic radiation.
* Has received a live-virus vaccination within 30 days of planned treatment start. Seasonal flu vaccines that do not contain live virus are permitted.
* Has allogenic haemopoietic stem cell (HSC) transplant.
* Prior treatment with idelalisib (a PI3K inhibitor).
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) >2.
* Poor bone marrow reserve.
* Poor organ function.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 109 (Actual)
Dates: Start 2018-02-21 (Actual); Primary Completion 2023-04-05 (Actual); Study Completion 2023-04-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (30):
- United States (4):
  - University of Colorado-Site Number:8400001, Denver, Colorado
  - University of Kansas Medical Center-Site Number:8400003, Kansas City, Kansas
  - Memorial Sloan-Kettering Cancer Center-Site Number:8400002, New York, New York
  - Fox Chase Cancer Center-Site Number:8400004, Philadelphia, Pennsylvania
- Australia (3):
  - Investigational Site Number :0360003, Wollongong, New South Wales
  - Investigational Site Number :0360002, Richmond, Victoria
  - Investigational Site Number :0360001, West Perth, Western Australia
- Brazil (3):
  - Investigational Site Number :0760003, Goiânia, Goiás
  - Investigational Site Number :0760001, Porto Alegre, Rio Grande do Sul
  - Investigational Site Number :0760004, São Paulo, São Paulo
- Canada (3):
  - Investigational Site Number :1240001, Montreal, Quebec
  - Investigational Site Number :1240005, Montreal, Quebec
  - Investigational Site Number :1240003, Sherbrooke, Quebec
- Czechia (3):
  - Investigational Site Number :2030002, Brno
  - Investigational Site Number :2030003, Ostrava - Poruba
  - Investigational Site Number :2030001, Prague
- France (4):
  - Investigational Site Number :2500004, Lille
  - Investigational Site Number :2500002, Nantes
  - Investigational Site Number :2500003, Pierre-Bénite
  - Investigational Site Number :2500001, Villejuif
- Investigational Site Number :3000001, Athens, Greece
- Investigational Site Number :3480002, Budapest, Hungary
- Italy (3):
  - Investigational Site Number :3800005, Rozzano, Milano
  - Investigational Site Number :3800003, Brescia
  - Investigational Site Number :3800001, Torino
- Spain (5):
  - Investigational Site Number :7240003, Barcelona, Barcelona [Barcelona]
  - Investigational Site Number :7240004, Badalona, Catalunya [Cataluña]
  - Investigational Site Number :7240002, Barcelona, Catalunya [Cataluña]
  - Investigational Site Number :7240005, Valencia, Valenciana, Comunidad
  - Investigational Site Number :7240006, Madrid

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were screened at 30 sites. The study was conducted i.e. participants were randomized at 29 sites in 10 countries. A total of 3 participants in Phase 1 and 106 participants in Phase 2 were enrolled (Phase 1)/randomized (Phase 2) from 21 Feb 2018 to 20 Mar 2019.
Pre-assignment Details: The study consisted of 2 phases: Phase 1 confirmed the feasibility of isatuximab/cemiplimab combination and Phase 2 further evaluated safety, efficacy and pharmacokinetics (PK) of combination versus isatuximab monotherapy. Participants in Phase 2 were randomized in a 1:1:1 ratio to receive either isatuximab monotherapy or combination therapy. The duration of study for a participant included a screening period (up to 21 days) and 3-month post treatment follow-up. Each cycle duration was 28 days.
Groups:
- Phase 1: Isatuximab + Cemiplimab Once Every 2 Weeks (Q2W): Participants received isatuximab 10 milligram/ kilogram (mg/kg) intravenous (IV) infusion once weekly for 4 weeks (QWx4) followed by Q2W (on Days 1, 8, 15 and 22 in Cycle 1, and on Days 1 and 15 in Cycle 2 and beyond of a 28-day cycle) and cemiplimab 250 mg IV infusion Q2W (on Days 1 and 15 every cycle of a 28-day cycle) until disease progression, unacceptable adverse events (AEs), consent withdrawal, or any other reason.
- Phase 2: Isatuximab: Participants received isatuximab 10 mg/kg IV infusion QWx4 followed by Q2W (on Days 1, 8, 15 and 22 in Cycle 1, and on Days 1 and 15 in Cycle 2 and beyond of a 28-day cycle) until disease progression, unacceptable AEs, consent withdrawal, or any other reason.
- Phase 2: Isatuximab + CemiplimabQ2W: Participants received isatuximab 10 mg/kg IV infusion QWx4 followed by Q2W (on Days 1, 8, 15 and 22 in Cycle 1, and on Days 1 and 15 in Cycle 2 and beyond of a 28-day cycle) and cemiplimab 250 mg IV infusion Q2W (on Days 1 and 15 every cycle of a 28-day cycle) until disease progression, unacceptable AEs, consent withdrawal, or any other reason.
- Phase 2: Isatuximab + Cemiplimab Once Every 4 Weeks (Q4W): Participants isatuximab 10 mg/kg IV infusion QWx4 followed by Q2W (on Days 1, 8, 15 and 22 in Cycle 1, and on Days 1 and 15 in Cycle 2 and beyond of a 28-day cycle) and cemiplimab 250 mg IV infusion Q4W (on Day 1 every cycle of a 28-day cycle) until disease progression, unacceptable AEs, consent withdrawal, or any other reason.
Period: Overall Study
Arm/Group | Phase 1: Isatuximab + Cemiplimab Once Every 2 Weeks (Q2W) | Phase 2: Isatuximab | Phase 2: Isatuximab + CemiplimabQ2W | Phase 2: Isatuximab + Cemiplimab Once Every 4 Weeks (Q4W)
Started (Enrolled for Phase 1; randomized for Phase 2) | 3 | 34 | 36 | 36
Randomized and Treated (Enrolled for Phase1; randomized for Phase 2. Phase 2 Isatuximab + CemiplimabQ2W, one participant was randomized but not treated.) | 3 | 34 | 35 | 36
Completed (Participants with end of study or death from any cause forms completed.) | 3 | 34 | 35 | 36
Not Completed | 0 | 0 | 1 | 0
Not completed — Incorrect completion of end of study form | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Phase 1:The Safety population: All screened participants who received at least 1 dose or a part of a dose of study treatments (isatuximab or cemiplimab), regardless of the amount of treatment administered. Phase 2: The Randomized population: All participants who gave informed consent, were assigned randomization number by interactive response technology (IRT), regardless of whether they received any study treatment or received a different study treatment from which they were randomized.
Groups:
- Phase 1: Isatuximab + CemiplimabQ2W: Participants received isatuximab 10 mg/kg IV infusion QWx4 followed by Q2W (on Days 1, 8, 15 and 22 in Cycle 1, and on Days 1 and 15 in Cycle 2 and beyond of a 28-day cycle) and cemiplimab 250 mg IV infusion Q2W (on Days 1 and 15 in all cycles every cycle of a 28-day cycle) until disease progression, unacceptable AEs, consent withdrawal, or any other reason.
- Phase 2: Isatuximab + CemiplimabQ4W: Participants isatuximab 10 mg/kg IV infusion QWx4 followed by Q2W (on Days 1, 8, 15 and 22 in Cycle 1, and on Days 1 and 15 in Cycle 2 and beyond of a 28-day cycle) and cemiplimab 250 mg IV infusion Q4W (on Day 1 every cycle of a 28-day cycle) until disease progression, unacceptable AEs, consent withdrawal, or any other reason.
- Total: Total of all reporting groups
Arm/Group | Phase 1: Isatuximab + CemiplimabQ2W | Phase 2: Isatuximab | Phase 2: Isatuximab + CemiplimabQ2W | Phase 2: Isatuximab + CemiplimabQ4W | Total
Number analyzed (Participants) | 3 | 34 | 36 | 36 | 109
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.7 (2.9) | 66.1 (9.3) | 63.7 (10.0) | 66.4 (9.2) | 65.4 (9.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 16 | 14 | 16 | 47
  Male | 2 | 18 | 22 | 20 | 62
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 2 | 3 | 3 | 8
  White | 3 | 29 | 30 | 29 | 91
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 3 | 3 | 3 | 9

OUTCOME MEASURES:

1. Primary Outcome: Phase 1: Number of Participants With Dose-Limiting Toxicities (DLTs)
Description: Potential DLTs were defined as the occurrence of any of the following adverse reactions at first treatment cycle, unless due to disease progression or obviously unrelated cause: Hematological DLTs: Grade(G) 4 neutropenia (N) for more than 7 consecutive days, G3 to G4 N complicated by fever (temperature greater than or equal to [>=] 38.5 degree Celsius on more than 1 occasion) or microbiologically/radiographically documented infection, G3 to G4 thrombocytopenia associated with clinically significant bleeding requiring clinical intervention or Non-hematological DLTs: G4 non-hematologic AE, G>=2 uveitis, G3 non-hematological AE lasting greater than (>)3 days despite optimal care support, delay in initiation of Cycle 2 >14 days due to treatment related laboratory abnormalities/AE. Any other AE that the investigator/study committee deemed to be dose-limiting, regardless of grade, was also considered as DLT.
Time Frame: Cycle 1 Day 1 to Day 28
Population: The DLT evaluable population consisted of participants in Phase 1 who received the planned doses of isatuximab and cemiplimab during Cycle 1, and who completed the DLT observation period of Cycle 1 after the first study treatment administration, unless they discontinued the study treatment(s) due to DLT.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1: Isatuximab + CemiplimabQ2W
Number analyzed (Participants) | 3
Participants | 0

2. Primary Outcome: Phase 1 and Phase 2: Number of Participants With Treatment-Emergent Adverse Events (TEAEs) and Treatment-Emergent Serious Adverse Events (TESAEs)
Description: An AE was defined as any untoward medical occurrence in a participant or clinical investigation participant administered with a pharmaceutical product and which did not necessarily have a causal relationship with study treatment. SAEs were any untoward medical occurrence that at any dose: resulted in death, was life-threatening, required inpatient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity, was a congenital anomaly/birth defect, was a medically important event. TEAEs were defined as an AE which occurred after the first dose of study treatment administration up to 30 days after the last dose of study treatment administration. The DLT observation period was 1 cycle (28 days). However, all AEs during treatment, unless due to disease progression or an obviously unrelated cause, were taken into consideration by the Study Committee for the determination of the maximum tolerated dose and recommended Phase 2 dose.
Time Frame: TEAEs were collected from the first dose up to 30 days after the last dose of study treatment, approximately 50 months
Population: Analysis was performed on the Safety population (tabulated according to treatment actually received [as treated]). There were 2 participants randomized in group isatuximab and isatuximab + cemiplimabQ4W respectively and who took another treatment/schedule.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1: Isatuximab + CemiplimabQ2W | Phase 2: Isatuximab | Phase 2: Isatuximab + CemiplimabQ2W | Phase 2: Isatuximab + CemiplimabQ4W
Number analyzed (Participants) | 3 | 33 | 37 | 35
Participants
  TEAEs | 3 | 33 | 36 | 33
  TESAEs | 1 | 17 | 17 | 21

3. Primary Outcome: Phase 2: Percentage of Participants With Overall Response Rate (ORR)
Description: ORR by Investigator using international myeloma working group (IMWG) response criteria:percentage of participants with complete response (CR) (including stringent CR [sCR]very good partial response [VGPR] and partial response [PR]).CR:negative immunofixation on serum and urine,disappearance of any soft tissue plasmacytomas,less than (<)5% plasma cells in bone marrow (BM) aspirates and normal free light chain(FLC)ratio (0.26-1.65).sCR:CR plus no clonal cells in BM biopsy.VGPR:serum and urine M-protein detectable by immunofixation,not electrophoresis;>=90% reduction in serum M-protein plus urine M-protein level<100mg/24hour(h);FLC only:>=90% decrease in difference between involved and uninvolved FLC levels.PR:>=50% reduction of serum M-protein and reduction in 24h urine M-protein by >=90% or <200mg/24h.In addition to above, if present at baseline,>=50% reduction in size (sum of products of maximal perpendicular diameters of measured lesions [SPD]) of soft tissue plasmacytomas required.
Time Frame: From Cycle 1 Day 1 up to primary analysis completion date of 9 Oct 2019 i.e., up to approximately 17 months
Population: The Randomized population consisted of all participants from Phase 2 who gave their informed consent and were assigned a randomization number by the IRT, regardless of whether participants received any study treatment or received a different study treatment from which they were randomized.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase 2: Isatuximab | Phase 2: Isatuximab + CemiplimabQ2W | Phase 2: Isatuximab + CemiplimabQ4W
Number analyzed (Participants) | 34 | 36 | 36
percentage of participants | 11.8 [3.30 to 27.45] | 25.0 [12.12 to 42.20] | 22.2 [10.12 to 39.15]

4. Secondary Outcome: Phase 2: Percentage of Participants With Clinical Benefit Rate (CBR)
Description: CBR by Investigator using IMWG response criteria: percentage of participants with CR (including sCR), VGPR, PR (all defined in previous OM) or MR. MR was defined as >= 25% but <= 49% reduction in serum M-protein and reduction in 24h urine M-protein by 50-89%, which still exceeded 200 mg/24h; if present at baseline, >=50% reduction in size (SPD) of soft tissue plasmacytomas was also required.
Time Frame: From Cycle 1 Day 1 up to primary analysis completion date of 9 Oct 2019 i.e., up to approximately 17 months
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase 2: Isatuximab | Phase 2: Isatuximab + CemiplimabQ2W | Phase 2: Isatuximab + CemiplimabQ4W
Number analyzed (Participants) | 34 | 36 | 36
percentage of participants | 23.5 [10.75 to 41.17] | 36.1 [20.82 to 53.78] | 38.9 [23.14 to 56.54]

5. Secondary Outcome: Phase 2: Duration of Follow-up
Description: Duration of follow-up was defined as the date of randomization to the date of last contact or death, whichever came first. Median duration of follow-up is reported.
Time Frame: From the date of randomization up to primary analysis completion date of 9 Oct 2019 i.e., up to approximately 17 months
Population: as for outcome 3
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase 2: Isatuximab | Phase 2: Isatuximab + CemiplimabQ2W | Phase 2: Isatuximab + CemiplimabQ4W
Number analyzed (Participants) | 34 | 36 | 36
months | 10.28 [8.739 to 11.368] | 8.84 [8.016 to 11.072] | 9.03 [8.016 to 10.875]

6. Secondary Outcome: Phase 2: Duration of Response (DOR)
Description: DOR: Time from date of first response (>=PR) that was subsequently confirmed to date of first documented progressive disease (PD) or death.DOR was determined only for participants who achieved a response of PR or better.If progression or death not observed, participant was censored at date of last valid disease assessment not showing disease progression performed prior to initiating further anticancer treatment and analysis cut-off date.PD(IMWG criteria):increase of >=25% from lowest confirmed value in any 1 of following:serum M-protein (absolute increase>=0.5 gram/deciliter[g/dL]), serum M-protein increase>=1g/dL if lowest M component >=5g/dL; urine M-component (absolute increase >=200mg/24h),appearance of new lesion(s),>=50% increase from nadir in SPD of >1 lesion or >=50% increase in longest diameter of a previous lesion >1cm in short axis,>=50% increase in circulating plasma cells (minimum 200 cells/microliter[c/mcL]) if that was the only measure of disease. PR: as defined in OM3.
Time Frame: From Cycle 1 Day 1 up to primary analysis completion date of 9 Oct 2019 i.e., up to approximately 17 months
Population: The Randomized population consisted of all participants from Phase 2 who gave their informed consent and were assigned a randomization number by the IRT, regardless of whether participants received any study treatment or received a different study treatment from which they were randomized. Only responders were included in the analysis.
Measure: Median (Full Range); unit: months
Arm/Group | Phase 2: Isatuximab | Phase 2: Isatuximab + CemiplimabQ2W | Phase 2: Isatuximab + CemiplimabQ4W
Number analyzed (Participants) | 4 | 9 | 8
months | 5.6 [4 to 7] | 4.7 [3 to 12] | 5.7 [2 to 12]

7. Secondary Outcome: Phase 2: Time to Response (TTR)
Description: TTR was defined as the time from randomization to first response (PR or better) that was subsequently confirmed. PR as per IMWG criteria was defined as >=50% reduction of serum M-protein and reduction in 24 hours urinary M-protein by >=90% or to <200 mg/24 hours. In addition to the above listed criteria, if present at baseline, a >=50% reduction in the size SPD of soft tissue plasmacytomas was also required.
Time Frame: From Cycle 1 Day 1 up to primary analysis completion date of 9 Oct 2019 i.e., up to approximately 17 months
Population: as for outcome 6
Measure: Median (Full Range); unit: months
Arm/Group | Phase 2: Isatuximab | Phase 2: Isatuximab + CemiplimabQ2W | Phase 2: Isatuximab + CemiplimabQ4W
Number analyzed (Participants) | 4 | 9 | 8
months | 1.5 [1 to 2] | 1.0 [1 to 3] | 1.0 [1 to 4]

8. Secondary Outcome: Phase 2: Progression Free Survival (PFS)
Description: PFS: Time interval from the randomization date to the date of the first documented disease progression that is subsequently confirmed or the date of death due to any cause, whichever came first. If progression or death was not observed, participant was censored at date of last valid disease assessment not showing disease progression performed prior to initiation of a further anticancer treatment or the analysis cut-off date. Analysis was performed by Kaplan-Meier method. PD (IMWG) criteria: increase of >=25% from lowest confirmed value in any 1 of following: serum M-protein (absolute increase >=0.5g/dL), serum M-protein increase >=1g/dL if lowest M component was >=5g/dL; urine M-component (absolute increase >=200mg/24h), appearance of new lesion(s),>=50% increase from nadir in SPD of >1 lesion or >=50% increase in the longest diameter of a previous lesion >1 cm in short axis or >=50% increase in circulating plasma cells (minimum of 200 c/mcL) if that was the only measure of disease.
Time Frame: From Cycle 1 Day 1 up to primary analysis completion date of 9 Oct 2019 i.e., up to approximately 17 months
Population: as for outcome 3
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase 2: Isatuximab | Phase 2: Isatuximab + CemiplimabQ2W | Phase 2: Isatuximab + CemiplimabQ4W
Number analyzed (Participants) | 34 | 36 | 36
months | 2.89 [1.971 to 3.811] | 3.75 [1.971 to 5.881] | 3.02 [2.793 to 5.158]

9. Secondary Outcome: Phase 2: Overall Survival (OS)
Description: OS was defined as the time interval from the date of randomization to death from any cause. Participants without death prior to the analysis cut-off date were censored at the last date the participant was known to be alive or the cut-off date, whichever came first. The results provided below corresponds to descriptive OS information at the time of primary analysis completion date of 09 October 2019.
Time Frame: From Cycle 1 Day 1 up to primary analysis completion date of 9 Oct 2019 i.e., up to approximately 17 months
Population: as for outcome 3
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase 2: Isatuximab | Phase 2: Isatuximab + CemiplimabQ2W | Phase 2: Isatuximab + CemiplimabQ4W
Number analyzed (Participants) | 34 | 36 | 36
months | NA [7.622 to NA] — NA indicates due to the limited follow-up time, most of participants were still alive, so the median OS and upper limit of confidence interval (CI) was not reached. | NA [6.801 to NA] — NA indicates due to the limited follow-up time, most of participants were still alive, so the median OS and upper limit of CI was not reached. | 12.78 [7.392 to NA] — NA indicates due to the limited follow-up time, most of participants were still alive, so upper limit of CI was not reached.

10. Secondary Outcome: Phase 1 and 2: Plasma Concentration Observed at the End of IV Infusion (Ceoi) of Isatuximab Alone and in Combination With Cemiplimab
Description: Plasma samples were collected at specified timepoints and those non-impacted by the bioanalytical issue were used for evaluation of Ceoi. It was calculated using non-compartmental analysis (NCA) after the first administration in Cycle 1. The PK population was defined independently for isatuximab and cemiplimab and consisted of all participants from the all-treated (AT) population with at least 1 available concentration post-baseline (whatever the cycle and even if dosing was incomplete) with adequate documentation of dosing and sampling dates and times.
Time Frame: At end of infusion (EOI) on Cycle 1 Day 1
Population: Analysis was performed on the PK population. "Isatuximab + Cemiplimab" arm includes 3 and 27 participants from phase 1 and phase 2, respectively. Same dose of isatuximab was administered to all participants in phase 1 and phase 2 part of study in Isatuximab + Cemiplimab Q2W and Q4W arms. Hence PK analysis was combined for phase 1 and phase 2 Isatuximab + Cemiplimab Q2W and Q4W arms.
Measure: Mean (Standard Deviation); unit: microgram (mcg)/mL
Groups:
- Phase 1 and 2: Combination Arm: Isatuximab + Cemiplimab: All participants who received isatuximab in combination with cemiplimab were included in this arm.
Arm/Group | Phase 2: Isatuximab | Phase 1 and 2: Combination Arm: Isatuximab + Cemiplimab
Number analyzed (Participants) | 10 | 30
microgram (mcg)/mL | 255 (72.1) | 239 (67.7)

11. Secondary Outcome: Phase 1 and 2: Maximum Observed Concentration (Cmax) of Isatuximab Alone and in Combination With Cemiplimab
Description: Plasma samples were collected at specified timepoints and those non-impacted by the bioanalytical issue were used for evaluation of Cmax. It was calculated using NCA after the first administration in Cycle 1.
Time Frame: At start of infusion (SOI), EOI, EOI+4 hours, 72 hours and 168 hours on Day 1 of Cycle 1
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: mcg/mL
Arm/Group | Phase 2: Isatuximab | Phase 1 and 2: Combination Arm: Isatuximab + Cemiplimab
Number analyzed (Participants) | 10 | 30
mcg/mL | 264 (68.0) | 247 (65.9)

12. Secondary Outcome: Phase 1 and 2: Time to Reach Cmax (Tmax) of Isatuximab Alone and in Combination With Cemiplimab
Description: Plasma samples were collected at specified timepoints and those non-impacted by the bioanalytical issue were used for evaluation of tmax. It was calculated using NCA after the first administration in Cycle 1.
Time Frame: At SOI, EOI, EOI+4 hours, 72 hours and 168 hours on Day 1 of Cycle 1
Population: as for outcome 10
Measure: Median (Full Range); unit: hour
Arm/Group | Phase 2: Isatuximab | Phase 1 and 2: Combination Arm: Isatuximab + Cemiplimab
Number analyzed (Participants) | 10 | 30
hour | 5.56 [3.25 to 10.50] | 4.85 [2.58 to 13.70]

13. Secondary Outcome: Phase 1 and 2: Last Concentration Observed Above the Lower Limit of Quantitation (Clast) of Isatuximab Alone and in Combination With Cemiplimab
Description: Plasma samples were collected at specified timepoints and those non-impacted by the bioanalytical issue were used for evaluation of Clast. It was calculated using NCA after the first administration in Cycle 1.
Time Frame: At SOI, EOI, EOI+4 hours, 72 hours and 168 hours on Day 1 of Cycle 1
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: mcg/mL
Arm/Group | Phase 2: Isatuximab | Phase 1 and 2: Combination Arm: Isatuximab + Cemiplimab
Number analyzed (Participants) | 10 | 30
mcg/mL | 85.7 (44.9) | 64.1 (32.1)

14. Secondary Outcome: Phase 1 and 2: Time of Clast (Tlast) of Isatuximab Alone and in Combination With Cemiplimab
Description: Plasma samples were collected at specified timepoints and those non-impacted by the bioanalytical issue were used for evaluation of tlast. It was calculated using NCA after the first administration in Cycle 1.
Time Frame: At SOI, EOI, EOI+4 hours, 72 hours and 168 hours on Day 1 of Cycle 1
Population: as for outcome 10
Measure: Median (Full Range); unit: hour
Arm/Group | Phase 2: Isatuximab | Phase 1 and 2: Combination Arm: Isatuximab + Cemiplimab
Number analyzed (Participants) | 10 | 30
hour | 155.00 [72.40 to 169.00] | 165.00 [70.20 to 239.00]

15. Secondary Outcome: Phase 1 and 2: Area Under the Concentration Versus Time Curve (AUC) From Time Zero to Tlast (AUClast) of Isatuximab Alone and in Combination With Cemiplimab
Description: AUClast was defined as the area under the plasma concentration versus time curve from time 0 to real time tlast calculated using the trapezoidal method over the dosing interval after the first administration in Cycle 1.
Time Frame: At SOI, EOI, EOI+4 hours, 72 hours and 168 hours on Day 1 of Cycle 1
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: (mcg*hour)/mL
Arm/Group | Phase 2: Isatuximab | Phase 1 and 2: Combination Arm: Isatuximab + Cemiplimab
Number analyzed (Participants) | 10 | 30
(mcg*hour)/mL | 21000 (7220) | 20200 (6590)

16. Secondary Outcome: Phase 1 and 2: AUC From Time 0 to Week 1 (AUC1week) of Isatuximab Alone and in Combination With Cemiplimab
Description: AUC1week was defined as the area under the plasma concentration versus time curve from time 0 to 1 week post dose calculated using the trapezoidal method over the dosing interval after the first administration in Cycle 1.
Time Frame: At SOI, EOI, EOI+4 hours, 72 hours and 168 hours on Day 1 of Cycle 1
Population: Analysis was performed on the PK population. "Isatuximab + Cemiplimab" arm includes 3 and 27 participants from phase 1 and phase 2, respectively. Same dose of isatuximab was administered to all participants in phase 1 and phase 2 part of study in Isatuximab + Cemiplimab Q2W and Q4W arms. Hence PK analysis was combined for phase 1 and phase 2 Isatuximab + Cemiplimab Q2W and Q4W arms. Only those participants with data available were analyzed.
Measure: Mean (Standard Deviation); unit: (mcg*hour)/mL
Arm/Group | Phase 2: Isatuximab | Phase 1 and 2: Combination Arm: Isatuximab + Cemiplimab
Number analyzed (Participants) | 10 | 29
(mcg*hour)/mL | 23000 (7250) | 21100 (6450)

17. Secondary Outcome: Phase 1 and 2: Number of Participants With Anti-Drug Antibodies (ADA) to Isatuximab
Description: ADA responses were categorized as treatment-induced ADA and treatment boosted ADA. Pre-existing ADA was defined as ADA that were present in samples drawn during the pre-treatment period. Treatment-induced ADA was defined as ADA that developed at any time during the ADA on-study observation period in participants without pre-existing ADA. Treatment boosted ADA was defined as pre-existing ADAs with a significant increase in the ADA titer during the study compared to the Baseline titer. The ADA evaluable population was defined independently for isatuximab and cemiplimab and consisted of all participants from AT population with at least 1 ADA result (negative, positive, or inconclusive) post-baseline.
Time Frame: From Cycle 1 Day 1 up to primary analysis completion date of 9 Oct 2019 i.e., up to approximately 20 months
Population: Analysis was performed on the ADA evaluable population."Isatuximab + CemiplimabQ2W" arm includes 3 and 36 participants from phase 1 and phase 2, respectively. Same dose of isatuximab was administered to all participants in phase 1 and phase 2 part of study in Isatuximab + Cemiplimab Q2W arms. Hence analysis was combined for phase 1 and phase 2 Isatuximab + Cemiplimab Q2W arms.
Measure: Count of Participants; unit: Participants
Groups:
- Phase 1 and 2: Isatuximab + CemiplimabQ2W: Participants received isatuximab 10 mg/kg IV infusion QWx4 followed by Q2W (on Days 1, 8, 15 and 22 in Cycle 1, and on Days 1 and 15 in Cycle 2 and beyond of a 28-day cycle) and cemiplimab 250 mg IV infusion Q2W (on Days 1 and 15 every cycle of a 28-day cycle) until disease progression, unacceptable AEs, consent withdrawal, or any other reason.
Arm/Group | Phase 2: Isatuximab | Phase 1 and 2: Isatuximab + CemiplimabQ2W | Phase 2: Isatuximab + CemiplimabQ4W
Number analyzed (Participants) | 32 | 39 | 34
Participants
  Pre-existing ADA | 0 | 1 | 0
  Treatment-induced | 0 | 0 | 0
  Treatment boosted | 0 | 0 | 0

18. Secondary Outcome: Phase 1 and 2: Number of Participants With ADA to Cemiplimab
Description: ADA responses were categorized as treatment-induced ADA and treatment boosted ADA. Pre-existing ADA was defined as ADA that were present in samples drawn during the pre-treatment period. Treatment-induced ADA was defined as ADA that developed at any time during the ADA on-study observation period in participants without pre-existing ADA. Treatment boosted ADA was defined as pre-existing ADAs with a significant increase in the ADA titer during the study compared to the Baseline titer.
Time Frame: From Cycle 1 Day 1 up to primary analysis completion date of 9 Oct 2019 i.e., up to approximately 20 months
Population: Analysis was performed on the ADA evaluable population. "Isatuximab + CemiplimabQ2W" arm includes 3 and 36 participants from phase 1 and phase 2, respectively. Same dose of isatuximab was administered to all participants in phase 1 and phase 2 part of study in Isatuximab + Cemiplimab Q2W arms. Hence analysis was combined for phase 1 and phase 2 Isatuximab + Cemiplimab Q2W arms.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1 and 2: Isatuximab + CemiplimabQ2W | Phase 2: Isatuximab + CemiplimabQ4W
Number analyzed (Participants) | 39 | 34
Participants
  Pre-existing ADA | 1 | 0
  Treatment-induced | 2 | 0
  Treatment boosted | 0 | 0

ADVERSE EVENTS:
Time Frame: TEAEs were collected from the first dose up to 30 days after the last dose of study treatment, approximately 50 months. All-Cause Mortality was reported for the whole study duration, approximately 62 months
Description: Analysis was performed on the Safety population (tabulated according to treatment actually received [as treated]). There were 2 participants randomized in group isatuximab and isatuximab + cemiplimabQ4W respectively and who took another treatment/schedule.
Groups:
- Phase 1: Isatuximab+Cemiplimab Q2W: Participants received isatuximab 10 mg/kg IV infusion QWx4 followed by Q2W (on Days 1, 8, 15 and 22 in Cycle 1, and on Days 1 and 15 in Cycle 2 and beyond of a 28-day cycle) and cemiplimab 250 mg IV infusion Q2W (on Days 1 and 15 in all cycles every cycle of a 28-day cycle) until disease progression, unacceptable AEs, consent withdrawal, or any other reason.
- Phase 2:Isatuximab + CemiplimabQ4W: Participants isatuximab 10 mg/kg IV infusion QWx4 followed by Q2W (on Days 1, 8, 15 and 22 in Cycle 1, and on Days 1 and 15 in Cycle 2 and beyond of a 28-day cycle) and cemiplimab 250 mg IV infusion Q4W (on Day 1 every cycle of a 28-day cycle) until disease progression, unacceptable AEs, consent withdrawal, or any other reason.
Arm/Group | Phase 1: Isatuximab+Cemiplimab Q2W | Phase 2: Isatuximab | Phase 2: Isatuximab + CemiplimabQ2W | Phase 2:Isatuximab + CemiplimabQ4W
All-Cause Mortality (participants affected / at risk) | 1/3 | 20/33 | 23/37 | 22/35
Serious Adverse Events (participants affected / at risk) | 1/3 | 17/33 | 17/37 | 21/35
Other Adverse Events (participants affected / at risk) | 3/3 | 31/33 | 34/37 | 27/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1: Isatuximab+Cemiplimab Q2W (N=3) | Phase 2: Isatuximab (N=33) | Phase 2: Isatuximab + CemiplimabQ2W (N=37) | Phase 2:Isatuximab + CemiplimabQ4W (N=35)
Covid-19 Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Catheter Site Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Encephalitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Encephalomyelitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Escherichia Bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Herpes Zoster Disseminated (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Lower Respiratory Tract Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Osteomyelitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Parainfluenzae Virus Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 2 (2) | 1 (1) | 5 (5)
Pneumonia Staphylococcal (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pulmonary Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Pyelonephritis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Respiratory Tract Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Salmonellosis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Septic Shock (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Upper Respiratory Tract Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Cancer Pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Colon Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neuroendocrine Carcinoma Of The Skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperviscosity Syndrome (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 2 (3) | 0 (0)
Tumour Lysis Syndrome (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Delirium (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Psychomotor Hyperactivity (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Radicular Pain (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Spinal Cord Compression (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cardiac Failure Congestive (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute Abdomen (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anal Haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Obstruction Gastric (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Small Intestinal Obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Bone Lesion (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bone Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pathological Fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acute Kidney Injury (Renal and urinary disorders) | 0 (0) | 3 (3) | 2 (2) | 2 (2)
Fanconi Syndrome Acquired (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haematuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Proteinuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Renal Failure (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary Tract Obstruction (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Disease Progression (General disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Multiple Organ Dysfunction Syndrome (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Non-Cardiac Chest Pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Platelet Count Decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Infusion Related Reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Euthanasia (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1: Isatuximab+Cemiplimab Q2W (N=3) | Phase 2: Isatuximab (N=33) | Phase 2: Isatuximab + CemiplimabQ2W (N=37) | Phase 2:Isatuximab + CemiplimabQ4W (N=35)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 3 (3) | 5 (5)
Labyrinthitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 2 (4)
Oral Candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Pneumonia (Infections and infestations) | 1 (1) | 1 (1) | 2 (2) | 2 (2)
Respiratory Tract Infection (Infections and infestations) | 0 (0) | 3 (4) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0) | 3 (3) | 0 (0)
Upper Respiratory Tract Infection (Infections and infestations) | 1 (2) | 4 (4) | 4 (9) | 7 (13)
Urinary Tract Infection (Infections and infestations) | 0 (0) | 3 (4) | 2 (3) | 3 (3)
Viral Upper Respiratory Tract Infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (1) | 3 (8)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 2 (2) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 4 (6) | 3 (3)
Decreased Appetite (Metabolism and nutrition disorders) | 1 (1) | 3 (3) | 4 (4) | 2 (3)
Agitation (Psychiatric disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 3 (4) | 0 (0)
Confusional State (Psychiatric disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 3 (3) | 2 (2) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Headache (Nervous system disorders) | 0 (0) | 3 (3) | 3 (5) | 4 (4)
Lethargy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neuralgia (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Peripheral Sensory Neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Hypertension (Vascular disorders) | 0 (0) | 3 (4) | 3 (3) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 5 (6) | 5 (7) | 2 (2)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Dyspnoea Exertional (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 1 (1) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (1) | 2 (4)
Abdominal Pain Upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 6 (8) | 7 (10) | 7 (10)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gingival Pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lip Oedema (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 5 (5) | 5 (7) | 5 (6)
Oral Papule (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 3 (3) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 2 (4) | 1 (1) | 6 (6)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 2 (2) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 5 (5) | 4 (6) | 2 (3)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3) | 7 (9) | 3 (3)
Bone Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 4 (4) | 3 (3) | 3 (3)
Groin Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (3) | 2 (2)
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 3 (5) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 4 (4) | 1 (1)
Neck Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 4 (4) | 2 (2) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Asthenia (General disorders) | 0 (0) | 3 (6) | 5 (5) | 2 (2)
Chills (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Disease Progression (General disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Fatigue (General disorders) | 0 (0) | 3 (3) | 8 (12) | 5 (5)
Influenza Like Illness (General disorders) | 0 (0) | 2 (2) | 1 (2) | 0 (0)
Oedema Peripheral (General disorders) | 1 (1) | 2 (2) | 1 (1) | 3 (4)
Pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 4 (7) | 6 (10) | 2 (3)
Weight Decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 4 (4)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 3 (3) | 1 (1) | 2 (2)
Infusion Related Reaction (Injury, poisoning and procedural complications) | 2 (2) | 18 (22) | 15 (15) | 15 (15)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor supports publication of clinical trial results but may request that investigators temporarily delay or alter publications in order to protect proprietary information. The Sponsor may also require that the results of multicenter studies be published only in their entirety and not as individual site data.

DOCUMENTS (2):
  • Study Protocol (2022-03-21): https://cdn.clinicaltrials.gov/large-docs/67/NCT03194867/Prot_000.pdf
  • Statistical Analysis Plan (2019-03-05): https://cdn.clinicaltrials.gov/large-docs/67/NCT03194867/SAP_001.pdf